CLINICAL TRIAL: NCT03220568
Title: Adipose Tissue Content of Fatty Acids Present in Dairy Fat and Risk of Stroke. The Danish Diet, Cancer and Health Cohort
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: KKH-AT
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subcutaneous adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fatty acids present in adipose tissue samples

SUMMARY:
Background: Although low-fat dairy products are an integral part of a diet recommended for stroke prevention, the role of dairy fat in relation to the risk of stroke is not yet clear.

Objective: Therefore the association of adipose tissue content of fatty acids, for which dairy products are a major source (12:0, 14:0, 14:1 cis-9, 15:0, 17:0, 18:1 trans-11 and 18:2 cis-9, trans-11), with incident total stroke and stroke subtypes will be investigated.

Design: The study is a case-cohort study nested within the Danish Diet, Cancer and Health cohort, including all incident stroke cases and a random sample of the total cohort.The fatty acid composition of adipose tissue biopsies was determined by gas chromatography and the content of specific fatty acids was expressed as percentage of total fatty acids. Stroke cases were identified in the Danish National Patient Registry and the diagnoses were individually verified. Cox proportional hazard regression will be used to estimate the association between fatty acids and stroke.

ELIGIBILITY:
Inclusion Criteria: Born in Denmark, aged 50-64 years, residing in the urban and suburban areas of Copenhagen and Aarhus, Denmark.

-

Exclusion Criteria: Pre-existing cancer diagnosis. Previous stroke.

-

Ages: 50 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Between 1993 and 1997, a total of 57,053 men and women were recruited. At the time of invitation, they were 50 to 64 years old, born in Denmark, residing in the urban and suburban areas of Copenhagen and Aarhus and had not been registered with a cancer diagnosis in the Danish Cancer Registry.
Sampling Method: Non-Probability Sample
Enrollment: 57053 (Actual)
Dates: Start 1993-11-24 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

PRIMARY OUTCOMES:
Stroke, including validated subtypes | From baseline until 30 November 2009